CLINICAL TRIAL: NCT06234475
Title: A Randomized 2 by 2 Factorial Trial on mHealth Support and Financial Incentives to Promote Smoking Cessation in Deprived Older Smokers
Brief Title: Smoking Cessation Program for the Older Smokers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: University Grants Committee, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Prof. Wang Man-Ping, Professor, The University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: SCFO
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cessation; Aged; Telemedicine; Motivation
Keywords: Smoking Cessation; Low-income older smokers; Mobile health; Incentive; Real-time personalized support; Factorial study
MeSH Terms: conditions — Smoking Cessation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mobile health group (Experimental): Smartphone mHealth support for smoking cessation by scheduled age-friendly multimedia e-messages and real-time personalized behavioral supports for 3 months.
  Interventions: Behavioral: Mobile health support
- Financial incentive group (Experimental): An escalating incentive scheme for smoking abstinence: HK$500 for using any SC services within 6 months, and HK$1000, 1500 and 2000 for biochemically validated abstinence at 3-, 6- and 12-month, respectively.
  Interventions: Behavioral: Financial incentive
- Combined intervention group (Experimental): Smartphone mHealth support for smoking cessation by scheduled age-friendly multimedia e-messages and real-time personalized behavioral supports for 3 months and an escalating incentive scheme for smoking abstinence: HK$500 for using any SC services within 6 months, and HK$1000, 1500 and 2000 for biochemically validated abstinence at 3-, 6- and 12-month, respectively.
  Interventions: Behavioral: Combine intervention
- Control group (Active Comparator): Brief advice
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Mobile health support — 1. Brief smoking cessation advice
  2. Health warning leaflet
  3. Smoking cessation information booklet
  4. Referral card
  5. E-messages on SC-related information and details on community SC services for 3 months
  6. Acceptance and Commitment Therapy based real-time Chat-based support for 3 months
  Arms: Mobile health group
Behavioral: Financial incentive — 1. Brief smoking cessation advice
  2. Health warning leaflet
  3. Smoking cessation information booklet
  4. Referral card
  5. An escalating incentive scheme for smoking abstinence: HK$500 for using any SC services within 6 months, and HK$1000, 1500 and 2000 for biochemically validated abstinence at 3-, 6- and 12-month, respectively.
  Arms: Financial incentive group
Behavioral: Combine intervention — 1. Brief smoking cessation advice
  2. Health warning leaflet
  3. Smoking cessation information booklet
  4. Referral card
  5. E-messages on SC-related information and details on community SC services for 3 months
  6. Acceptance and Commitment Therapy based real-time Chat-based support for 3 months
  7. An escalating incentive scheme for smoking abstinence: HK$500 for using any SC services within 6 months, and HK$1000, 1500 and 2000 for biochemically validated abstinence at 3-, 6- and 12-month, respectively.
  Arms: Combined intervention group
Behavioral: Control group — 1. Brief smoking cessation advice
  2. Health warning leaflet
  3. Smoking cessation information booklet
  4. Referral card
  5. E-messages on SC-related information and details on community SC services for 3 months for those without abstinence at 12-month follow-up after follow-ups ending
  6. Acceptance and Commitment Therapy based rear-time Chat-based support for 3 months for those without abstinence at 12-month follow-up after follow-ups ending
  Arms: Control group

SUMMARY:
This study aims to assess the effect of mobile health (mHealth) support or financial incentives and their interactive intervention effect on smoking cessation (SC) in old smokers in Hong Kong (HK).

DETAILED DESCRIPTION:
Low-income older smokers are disproportionally harmed by tobacco use and the evidence of effectiveness of smoking cessation (SC) intervention for this deprived group is scarce. Leveraging evidence of effectiveness of mHealth support and financial incentives in other adults, the investigators propose a scalable mHealth and/or financial incentives model using age-friendly components for the deprived older smokers.

The 2x2 factorial design consists of 2 interventions, including (1) smartphone mHealth support by scheduled age-friendly multimedia e-messages and real-time personalized behavioral supports for 3 months, and (2) an escalating incentive scheme for smoking abstinence: HK$500 for using any SC services within 6 months, and HK$1000, 1500 and 2000 for biochemically validated abstinence at 3-, 6- and 12-month, respectively.

The study aims to assess the effectiveness of two interventions and their interactive intervention effect.

ELIGIBILITY:
Inclusion Criteria:

1. Smokers aged 60 years or above;
2. Currently smoking cigarettes or alternative tobacco products daily in the past 3 months with an exhaled carbon monoxide (CO) level ≥4ppm or salivary cotinine >30 ng/ml;
3. Have a mobile phone that can receive short message/messaging Service (SMS) or instant messages (IM);
4. Having a household monthly income lower than the median income of domestic household in Hong Kong

6. Hong Kong residents able to communicate in Chinese.

Exclusion Criteria:

1. Smokers not physically nor mentally fit for communication;
2. Smokers currently using SC services;
3. Hospitalized smokers;
4. Not having a mobile phone or perceived difficulty in using mobile phone or communication Apps

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The biochemically validated smoking abstinence | the 6-month follow-ups
  Smoking abstinence is defined by exhaled CO < 4 ppm and salivary cotinine <30 ng/ml

SECONDARY OUTCOMES:
The biochemically validated smoking abstinence | the 3- and 12-month follow-ups
  Smoking abstinence is defined by exhaled CO < 4 ppm and salivary cotinine <30 ng/ml
Self-reported 7-day point-prevalence abstinence | 3-, 6-, and 12-month follow-ups
  Smokers who did not smoke even a puff in the 7 days preceding the follow-up
Self-reported smoking change | 3-, 6-, and 12-month follow-ups
  Self-reported change in number of cigarettes smoked daily of at least less 50% of the baseline number
Self-reported self-efficacy of quitting | 3-, 6-, and 12-month follow-ups
  Self-reported self-efficacy of quitting includes the perception of quitting importance, difficulty and confidence, assessing by an item scaled with 0-10, respectively. The score of zero refers to very unimportant, very easy, or very unconfident. The score of 10 refers to very important, very difficult or very confident, respectively. Higher score refers to higher perception of quitting importance, difficulty and confidence.
Self-reported quit attempts | 3-, 6-, and 12-month follow-ups
  Self-reported quit attempt
Nicotine dependence level | 3-, 6-, and 12-month follow-ups
  Fagerstrom Test for Nicotine Dependence (FTND)
Smoking cessation services use | 3-, 6-, and 12-month follow-ups
  Using the smoking cessation service from hospitals or government in Hong Kong
Self-reported intention to quit | 3-, 6-, and 12-month follow-ups
  self-reported intention to quit in next days

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No